CLINICAL TRIAL: NCT01864109
Title: A Phase II Trial of Irinotecan and Temozolomide in Combination With Existing High Dose Alkylator Based Chemotherapy for Treatment of Patients With Newly Diagnosed Ewing Sarcoma
Brief Title: Irinotecan and Temozolomide in Combination With Existing High Dose Alkylator Based Chemotherapy for Treatment of Patients With Newly Diagnosed Ewing Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-068
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Newly Diagnosed Ewing Sarcoma
Keywords: CYCLOPHOSPHAMIDE (CYTOXAN); DOXORUBICIN/ADRIAMYCIN; ETOPOSIDE (VP-16); IFOSFAMIDE; IRINOTECAN (CPT-11) CAMPTOSAR; TEMOZOLOMIDE; VINCRISTINE; 13-068
MeSH Terms: interventions — Cyclophosphamide; Vincristine; Ifosfamide; Etoposide; Surgical Procedures, Operative; Radiotherapy; Temozolomide; Irinotecan; Mesna; Dexrazoxane; Granulocyte Colony-Stimulating Factor

ARMS (2):
- Patients with localized disease (Experimental): Patients with localized disease will receive six cycles of the combination as "maintenance" therapy following standard chemotherapy.
  * Cycles 4-6 will include:
    * Ifosfamide 2,800 mg/m2/day on days 1-5
    * Etoposide 100 mg/m2/day on days 1-5
  * Cycle 7 will include :
    * Cyclophosphamide will be given on days 1 and 2 at a dose of 2,100 mg/m2/day, or for patients < 10 years of age at a dose of 70 mg/kg/day
    * Doxorubicin will be given on days 1 and 2 at a dose of 37.5 mg/m2/day
    * Vincristine will be given on day 1 at a dose of 2 mg/m2 or 0.067 mg/kg (whichever is lower, to a max dose of 2 mg)
  * Cycles 8-13 will include:
    * Irinotecan will be given on 10 days over weeks 1 and 2 of a cycle at a dose of 20 mg/m2/day intravenously
    * Temozolomide will be given daily on the first 5 days of irinotecan administration at a dose of 100 mg/m2/day orally or intravenously
  Interventions: Drug: Cyclophosphamide; Device: Doxorubicin; Drug: Vincristine; Drug: Ifosfamide; Drug: Etoposide; Procedure: Surgery; Radiation: Radiation Therapy*; Drug: Temozolomide; Drug: Irinotecan; Drug: Mesna; Drug: Dexrazoxane; Drug: G-CSF
- Patients with metastatic disease (Experimental): Patients will get 10 cycles of the combination intercalated between the final 4 cycles of standard chemotherapy.
  * Cycles 4, 5, 7, 8, 10, 11, 13, 14, 16, and 17 will include:
    * Irinotecan will be given on 10 days over weeks 1 and 2 of a cycle at a dose of 20 mg/m2/day intravenously
    * Temozolomide will be given daily on the first 5 days of irinotecan administration at a dose of 100 mg/m2/day orally or intravenously
  * Cycles 6, 9, and 12 will include:
    * Ifosfamide 2,800 mg/m2/day on days 1-5
    * Etoposide 100 mg/m2/day on days 1-5
  * Cycle 15 will include:
    * Cyclophosphamide will be given on days 1 and 2 at a dose of 2,100 mg/m2/day, or for patients < 10 years of age at a dose of 70 mg/kg/day
    * Doxorubicin will be given on days 1 and 2 at a dose of 37.5 mg/m2/day
    * Vincristine will be given on day 1 at a dose of 2 mg/m2 or 0.067 mg/kg (whichever is lower, to a max dose of 2 mg)
  Interventions: Drug: Cyclophosphamide; Device: Doxorubicin; Drug: Vincristine; Drug: Ifosfamide; Drug: Etoposide; Procedure: Surgery; Radiation: Radiation Therapy*; Drug: Temozolomide; Drug: Irinotecan; Drug: Mesna; Drug: Dexrazoxane; Drug: G-CSF

INTERVENTIONS:
Drug: Cyclophosphamide
Device: Doxorubicin
Drug: Vincristine
Drug: Ifosfamide
Drug: Etoposide
Procedure: Surgery
Radiation: Radiation Therapy* — If local control includes RT, RT should be given concurrently with chemotherapy cycles
Drug: Temozolomide
Drug: Irinotecan
Drug: Mesna — Mesna 2,100 mg/m2 (or 70 mg/kg if < 10 yrs of age) administered intravenously in concordance with institutional pediatric administration guidelines.
Drug: Dexrazoxane — Dexrazoxane 375 mg/m2 intravenously over approximately 15-30 minutes and as clinically indicated. To be administered immediately prior to doxorubicin.
Drug: G-CSF — G-CSF-to be administered after the completion of appropriate chemotherapy cycles as per institutional guidelines.

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, the combination of irinotecan and temozolomide has on Ewing sarcoma.

Irinotecan and temozolomide are chemotherapy drugs that are used very often to treat pediatric patients at MSKCC. The investigators have used these two drugs for many years to treat patients with Ewing sarcoma whose cancer has relapsed.

For patients with newly diagnosed Ewing sarcoma the current standard of care at MSKCC is a five drug chemotherapy regimen in combination with surgery and/or radiation therapy. This standard regimen is called the EFT regimen. . Some patients with Ewing sarcoma do not have their cancer cured by the chemotherapy and surgery/radiation therapy.

This study adds the chemotherapy drugs called irinotecan and temozolomide to the standard EFT regimen. The investigators are trying to improve the success of standard therapy by adding these drugs. The use of irinotecan and temozolomide in this study is experimental because they have not been used before in patients with newly diagnosed Ewing sarcoma. However the investigators have found these drugs to be effective in patients with relapsed Ewing sarcoma. It is not known if adding these two drugs will improve the outcomes of patients treated for Ewing sarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to one year and less than or equal to 40 years at the time of diagnosis
* Newly diagnosed, previously untreated patients with histologically or molecularly confirmed Ewing sarcoma
* Adequate hematologic function:
* Absolute neutrophil count ≥ 1,000/K/mcl
* Platelet count ≥ 100,000/Kmcl
* Adequate renal function:
* Normal creatinine for age (See table below) OR
* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73 m2 Age(Years) Maximum Serum Creatinine (mg/dL) ≤ 5 0.8 6 to ≤ 10 1 11 to ≤ 15 1.2 ≥ 16 1.5

Adequate hepatic function:

* Total bilirubin ≤ 1.5 x the ULN
* AST ≤ 2.5 x the ULN [in the absence of hepatic involvement of tumor. Patients with hepatic involvement are considered eligibile for study]
* ALT ≤ 2.5 x the ULN [in the absence of hepatic involvement of tumor. Patients with hepatic involvement are considered eligibile for study]

Normal cardiac function:

* Shortening fraction ≥ 28% by echocardiogram OR
* Left ventricular ejection fraction (LVEF) ≥ 50% on technetium- 99m pertechnetate radionuclide cineangiography (MUGA) or echocardiogram
* Patients must consent to an indwelling central venous catheter.
* Sexually active patients of reproductive potential must be willing to use an effective method of contraception.

Exclusion Criteria:

* Prior chemotherapy or radiotherapy (other than limited, emergent radiotherapy for treatment of eg. spinal cord compromise or threatened airway)
* Pregnant or breastfeeding females

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 83 (Actual)
Dates: Start 2013-05; Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
event free survival of patients with localized disease | 4 years
  We will determine event free survival from the time of study entry for all patients. An event would include death from any cause, progression of tumor, recurrence of tumor, or second malignancy.
  Progressive disease (PD) will be defined according to RECIST 1.1.

SECONDARY OUTCOMES:
event free survival of patients with metastatic disease | 4 years
  We will determine event free survival from the time of study entry for all patients. An event would include death from any cause, progression of tumor, recurrence of tumor, or second malignancy.
  Progressive disease (PD) will be defined according to RECIST 1.1.
adverse event profile | 2 years
  Toxicities are graded by the Common Toxicity Criteria (Version 4.0) developed by the National Cancer Institute (NCI) of the USA.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Slotkin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Cancer Center Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/